CLINICAL TRIAL: NCT01100346
Title: A Prospective, Single Center, Observational Study on the Predictive Factors of Ovarian Response in Ovulation Induction (OI) With Intrauterine Insemination (IUI) of a Gonal-f Low-dose Step-up Regimen
Brief Title: Predictive Factors of Ovarian Response in Ovulation Induction With Intrauterine Insemination of a Gonal-f Low-dose Regimen
Status: Terminated | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Ltd., Taiwan (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 700623-509
Record Dates: First submitted 2010-03-10; First posted 2010-04-08 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2012-11

CONDITIONS: Infertility
Keywords: Ovulation induction; Intrauterine insemination; Gonal-f; Controlled ovarian stimulation; Infertility
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gonal-f (Follitropin alpha) — A starting dose of 75 IU/day subcutaneously is maintained for a period of 7 to 14 days. The follitropin alpha dose would be subsequently increased by 37.5 IU/day at weekly intervals based on the ovarian response.
  Other Names: Gonal-f

SUMMARY:
This is a single center, prospective, observational study on the use of Gonal-f in controlled ovarian hyperstimulation (COH) in subjects undergoing ovulation induction/ intrauterine insemination (OI/IUI) therapy across Taiwan. It has been observed in the previous studies that COH with follicle stimulating hormone (FSH) is considered as one of the positive predictors of an ongoing pregnancy. Many studies in the past have tried to predict the FSH threshold, defined as the FSH dose on the day when a follicle is >10 mm in diameter, but no studies have been conducted to date to determine the predictive factors for a monofollicular development after COH in IUI cycles. Monofollicular growth contributes significantly to the reduction of multiple pregnancies and thus minimize the risks associated with such pregnancies. This study would provide preliminary data on the factors associated with a monofollicular development in Gonal-f treated cycles using a low dose step-up regimen.

DETAILED DESCRIPTION:
Ovarian stimulation improves the cycle fecundity rate in part by increasing the number of follicles available for fertilisation and correcting subtle, unpredictable ovulatory dysfunction. Intrauterine insemination is an established treatment for subfertility due to cervical factors, male factors, or unexplained etiology. Ovulation induction aims at the selection of a single follicle that would be able to reach the pre-ovulatory size and rupture. The ovarian sensitivity to FSH (FSH threshold) has to be identified to avoid multiple follicular development and hence, the lowest effective dose of FSH should be used in treating infertility.

Treatment in subjects is individualised and is monitored by serum estradiol (E2) measurements and ultrasound scans of the ovaries to assess the endometrial thickness. It has been observed in earlier studies that in OI for unexplained non-conception, induction of more than one follicle did not improve the ongoing pregnancy rate but increased the risk of multiple pregnancies. Therefore, to reduce the number of multiple pregnancies, in all IUI cycles for unexplained non-conception, monofollicular growth was suggested.

The 'low-dose step-up' protocol is the most suitable method to establish an appropriate FSH threshold, which involves a starting FSH dose of 75 IU/day given for 7 to 14 days. Subsequent dose increments of 37.5 IU/day at weekly intervals is determined based on the ovarian response, usually when a follicle of diameter ≥10 mm is not seen in the ovaries. Human chorionic gonadotrophin (hCG) is then injected when the leading follicle is ≥18 mm in diameter.

OBJECTIVES

Primary objective:

* To describe the outcome of treatment in a cohort of subjects undergoing OI/IUI therapy using Gonal-f

Secondary objective:

* To explore the predictive factors of ovarian response in OI/IUI therapy using a low-dose step-up regimen

This study is planned to enrol 30 female subjects from 1 centre in Taiwan. Each subject can receive up to 3 treatment cycles. Before undergoing a controlled ovarian stimulation with Gonal-f, a thorough gynaecologic and endocrinologic evaluation of the subject will be performed and the subjects will be given the first administration of Gonal-f low dose step up regimen for the controlled ovarian stimulation at the baseline visit. The objective of the Gonal-f therapy is to develop a single mature graafian follicle from which the ovum will be liberated after the administration of hCG. If a subject fails to respond adequately after 4 weeks of treatment, the cycle will be abandoned and the subject would recommence the treatment at a higher starting dose than in the abandoned cycle. If an excessive response is obtained, treatment would be stopped and hCG administration will be withheld and in the next cycle the treatment would start at a dosage lower than that of the previous cycle. Each enrolled subject will be followed up until the confirmation of her pregnancy status.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged between 20 and 35 years
* Subjects with regular menstrual cycle of 25 - 35 days
* Subjects with both ovaries
* Subjects with normal uterine cavity as investigated by either ultrasound scan or hysteroscopy and patent fallopian tube
* Subjects with baseline serum FSH level within normal range of the clinic
* Subjects whose male partner's semen is considered adequate for IUI in accordance to the centre's standard practice

Exclusion Criteria:

* Subjects with any contraindication to being pregnant and/or carrying a pregnancy to term
* Subjects with extrauterine pregnancy or abortion in the past 3 months
* Subjects with abnormal gynaecological bleeding of undetermined origin
* Subjects with history of OHSS
* Subjects with known hypersensitivity to recombinant FSH preparations or any of their recipients

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female subjects with regular menstrual cycles aged between 20 and 35 years in Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Number of follicles 11-15 mm and ≥ 16 mm in diameter, estradiol (E2) levels and endometrial thickness | On the day of hCG administration (during 24-48 hrs after the last Gonal-f injection)
Total dose of Gonal-f used during stimulation, threshold of Gonal-f dose (daily dose of Gonal-f when follicular growth is > 11 mm in diameter)and duration of Gonal-f treatment | During the period of ovarian stimulation
Outcomes of the treatment (Pregnancy status) | Stimulation start to pregnancy assessment
  Clinical pregnancy, multiple pregnancy, miscarriage, cycle cancellation, Ovarian hyperstimulation syndrome (OHSS) and severity.

SECONDARY OUTCOMES:
Proportion of subjects with monofollicular development | On the day of hCG administration (during 24-48 hrs after the last Gonal-f injection)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Ltd., Taiwan
Locations (1):
- Far Eastern Memorial Hospital, No.21 Nan-Ya S. Rd., Sec.2 Pan-Chiao, Taipei, Taiwan